CLINICAL TRIAL: NCT04522388
Title: A Pilot Study Examining the Effect of Nutritional Supplementation on Skeletal Muscle Mass in Patients Awaiting Lung Transplant
Brief Title: Examining the Effect of Nutritional Supplementation on Skeletal Muscle Mass in Patients Awaiting Lung Transplant
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to lack of enrollment and sponsored funding for this project
Sponsor: Johns Hopkins University (Other)
Collaborators: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00228299
Record Dates: First submitted 2020-08-18; First posted 2020-08-21 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Lung Transplant; Complications
Keywords: pre-hab; nutrition

STUDY DESIGN:
Intervention Model Description: Ensure Enlive, Nutritional shake, twice a day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Nutritional shakes, Ensure Enlive, twice per day orally in patients awaiting lung transplant
  Interventions: Dietary Supplement: Ensure Enlive

INTERVENTIONS:
Dietary Supplement: Ensure Enlive — Ensure Enlive shake twice a day

SUMMARY:
This non-randomized pilot study aims to investigate whether a protein rich nutritional shake (Ensure Enlive) given to patients pre-transplant will decrease skeletal muscle loss (measured by quadriceps ultrasound) and improve nutritional state (measured by Nutritional Risk Index). A nutritional supplement would be a cost-effective solution to treat malnutrition, a known risk factor implicated in poor outcomes for lung transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years or older who are listed for single or double lung transplant
* Subject provides written informed consent to participate in this study

Exclusion Criteria:

* Subject with history of Galactosemia
* Subject with history of milk protein allergy
* Subject with history of soy protein allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
Effect of nutritional supplementation on skeletal muscle mass as assessed by ultrasound of the quadriceps | Pre-transplant
  To examine the effect of nutritional supplementation on skeletal muscle mass in patients with end stage lung disease who are awaiting lung transplant, measured by ultrasound of the quadriceps.

SECONDARY OUTCOMES:
Effect of nutritional supplementation on Nutritional Risk index as assessed by serum albumin level | Pre-transplant
  To examine the effect of nutritional supplementation on Nutritional Risk index, measured by serum albumin level.

CONTACTS AND LOCATIONS:
Overall Officials: Errol Bush, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will be
Supporting Information: CSR
Time Frame: Data will be available upon completion of the study analysis
Access Criteria: Upon request to principal investigator

REFERENCES:
- [Background] Hsu J, Krishnan A, Lin CT, Shah PD, Broderick SR, Higgins RSD, Merlo CA, Bush EL. Sarcopenia of the Psoas Muscles Is Associated With Poor Outcomes Following Lung Transplantation. Ann Thorac Surg. 2019 Apr;107(4):1082-1088. doi: 10.1016/j.athoracsur.2018.10.006. Epub 2018 Nov 14. PMID 30447192
- [Background] Chamogeorgakis T, Mason DP, Murthy SC, Thuita L, Raymond DP, Pettersson GB, Blackstone EH. Impact of nutritional state on lung transplant outcomes. J Heart Lung Transplant. 2013 Jul;32(7):693-700. doi: 10.1016/j.healun.2013.04.005. Epub 2013 May 9. PMID 23664761
- See also: Sarcopenia of the Psoas Muscles Is Associated With Poor Outcomes Following Lung Transplantation — https://www.ncbi.nlm.nih.gov/pubmed/30447192
- See also: Impact of nutritional state on lung transplant outcomes — https://www.ncbi.nlm.nih.gov/pubmed/23664761